CLINICAL TRIAL: NCT01337557
Title: Use of BEPREVE (Bepotastine Besilate Ophthalmic Solution) 1.5% for Allergic Conjunctivitis and Contact Lenses
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hom, Milton M., OD, FAAO (Individual)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: Milton M. Hom, OD, FAAO., Private Practice
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MAC-03-11
Record Dates: First submitted 2011-04-14; First posted 2011-04-19 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Allergic Conjunctivitis
Keywords: Allergic conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — bepotastine; bepotastine besilate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bepotastine (Experimental)
  Interventions: Drug: Bepotastine

INTERVENTIONS:
Drug: Bepotastine — 1.5% bid
  Other Names: Bepreve

SUMMARY:
The purpose of this study is to assess if BEPREVE (bepotastine besilate ophthalmic solution) 1.5% will have an effect on contact lens wear in patients with contact lens intolerance due to allergic conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* History of allergic conjunctivitis
* History of contact lens intolerance
* Between the ages of 18 and over inclusive.
* Males or females
* Patient is in generally good & stable overall health.
* Patient likely to comply with study guidelines & study visits. Informed consent signed.
* Are willing/able to return for all required study visits.
* Are willing/able to follow instructions from the study investigator and his/her staff.
* If a woman capable of becoming pregnant, agree to have urine pregnancy testing performed at screening (must be negative) and agree to use a medically acceptable form of birth control throughout the study duration and for at least one week prior to and after completion of the study. Women considered capable of becoming pregnant include all females who have experienced menarche and who have not experienced menopause (as defined by amenorrhea for greater than 12 consecutive months) or have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy).
* Have signed informed consent approved by Institutional Review Board or Independent Ethics Committee.

Exclusion Criteria:

* Corneal refractive surgery within 6 months of this study.
* Current use of Restasis
* Intra-ocular surgery within 6 months or ocular laser surgery within 6 months.
* Pregnant or lactating women.
* Ocular pathology (includes glaucoma and cataract), which could impact results and/or place patient at risk.
* Systemic or injected corticosteroids (including oral, parenteral, intravenous, rectal) 30 days;
* Nasal or inhaled or ocular corticosteroids 14 days;
* Nasal or inhaled ipratropium bromide (or atropine), inhaled nedocromil, or nasal, inhaled, or ophthalmic sodium cromolyn 14 days;
* Agents with antihistaminic/anticholinergic activity (e.g. antidepressants, antipsychotics) 14 days;
* Leukotriene pathway modifiers (Accolate, Singulair, Zyflo) 10 days;
* Ocular anti-allergy medications including lodoxamide (Alomide), olopatadine (Patanol/Pataday), emedastine difumarate (Emadine), epinastine (Elestat), levocabastine (Livostin) 7 days;
* Non-steroidal anti-inflammatory ophthalmics including bromfenac (Xibrom), ketorolac (Acular/Acuvail), nepafenac (Nevanac), flurbiprofen (Ocufen), suprofen (Profenal), diclofenac (Voltaren) 7 days;
* OTC ophthalmic decongestant, antihistamine, or decongestant/antihistamine combinations 3 days;
* Other anticholinergic agents 3 days
* Immunotherapy injection 1 day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2011-05; Primary Completion 2011-09 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Questionnaire | 8 weeks
  Contact lens comfort and wearing times (measured in hours)

CONTACTS AND LOCATIONS:
Overall Officials: Milton M Hom, OD FAAO, Principal Investigator — Private Practice